CLINICAL TRIAL: NCT02790385
Title: Use of Incisional Negative Pressure Wound Dressing Versus Standard Dry Gauze Dressing for Wound Closure in Patients Undergoing Spinal Surgery - A Multicentre Randomized Control Trial
Brief Title: Negative Pressure Wound Therapy - A Multi-Centered Randomized Control Trial
Acronym: NPWT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H13-03020
Record Dates: First submitted 2014-02-07; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: to See Whether Negative Pressure Wound Therapy Decreases Wound Infections.
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NPWT (Experimental): subjects will undergo negative pressure wound therapy
  Interventions: Device: Negative Pressure Wound Therapy
- Standard Gauze (Active Comparator): standard method of using gauze and dressing will be utilized
  Interventions: Other: Standard Gauze Treatment

INTERVENTIONS:
Device: Negative Pressure Wound Therapy
  Arms: NPWT
Other: Standard Gauze Treatment
  Arms: Standard Gauze

SUMMARY:
Children with neuromuscular disorders such as cerebral palsy, children with kyphosis and post-traumatic scoliosis have higher infection rates after scoliosis surgery than healthy children who undergo scoliosis surgery. The purpose of our study is to compare the effect of NPWT on infection rates when compared to standard gauze dressing. Participants will be randomized to the "NPWT" or "standard dressing" group. We will compare infection rates between the two groups. We hypothesize participants in the "NPWT" group will have a lower infection rate.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Consent/assent to participate in the study
* Undergoing posterior spinal surgery categorized as High-Risk for infection, defined as greater than 4% risk of deep or superficial infection based previous reported literature. Procedures qualifying for study are listed below:
* Kyphosis (any type)
* Posttraumatic Scoliosis
* Neuromuscular Scoliosis

Exclusion Criteria:

* Previous incisions over the operative site
* History of keloid formation
* Allergy to tape
* Does not consent/assent to participate in the study
* Previous or Active Spinal infection
* Dural tear
* Hemophiliac
* Two Stage procedure
* Unable to follow standard antibiotic protocols

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 870 (Estimated)
Dates: Start 2014-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Wound Infection | up to post op day 14
  Wounds will be classified as prolonged discharge if they have persistent sterile drainage on post-op day 5 or after, or as "infected," if cellulitis is found at suture line (erythema >1cm + tenderness + localized swelling + warmth). Wound assessment will be carried out by a clinical fellow on day 5 and subsequent days till discharge. Patients will also be assessed for other signs of infection such as Fever, Chills, and increase in pain or changes in appetite. Standard infection work-up will be utilized to rule in or rule out infection.

SECONDARY OUTCOMES:
Time for wound closure | intraoperatively
  This will be measured intra-operatively in the operating room from the beginning of deep wound closure till complete skin closure either with standard treatment or by NPWT. Though this outcome measure may not appear to have much value as these surgeries are of a long duration, we considered it important from the surgeon's perspective.
Cosmetic results | 12 weeks post op
  (Hollander wound evaluation scale): This is a validated cosmetic scoring system [8], which gives a score from 0 to 6. The score addresses six clinical variables: step off borders, contour irregularities, scar width, edge inversion, excessive inflammation, and overall cosmetic appearance. Each of these categories is graded on a 0- or 1-point scale where a score of 6 is considered optimal. At 12 weeks post-op follow-up, assessment of the scar will be carried out by an independent investigator who will be blinded to which treatment group the patient belongs to.
Caregiver/parental satisfaction | 12 weeks post op
  This will analyzed on a visual analog scale (VAS)
Wound dehiscence | psot op day 5 to discharge
  Any gaping of the spinal wound > 5cm exposing subcutaneous tissue or deeper planes will be considered as indicative of wound dehiscence. This will be looked for at the 5th post- operative day during dressing change till 14 days post-op.
Foreign body reaction | 12 weeks post op
  Any evidence of foreign body reaction will be looked for at the two week mark and at 12 weeks post-op follow up. The presence of swelling under the wound over the suture or NPWT site in the absence of fever, significant redness and tenderness will be indicative of foreign body reaction.

CONTACTS AND LOCATIONS:
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada